CLINICAL TRIAL: NCT02938390
Title: Ultrasound Localization of Intercostal Perforating Vessels Reduces Post-Operative Wound Complications From Nipple Sparing Mastectomy
Brief Title: Localization of Intercostal Perforating Vessels Reduces Wound Complications From Nipple Sparing Mastectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Amita Health (Other)
Responsible Party: Principal Investigator, Robert Maganini, MD, Principal Investigator, Amita Health
Other Study IDs: Nipple Sparing Study
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Nipple Sparing Mastectomy; Ultrasound
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ultrasound for localizing intercostal perforating vessels — Use of an Intra-operative ultrasound during nipple sparing mastectomy to localize intercostal perforating vessels.

SUMMARY:
Approximately 100 women scheduled for NSM will be consented pre-operatively to participate in the study. US will be performed after induction of general anesthesia, prior to surgery using Sonosite™ portable US, 5-12mHz transducer using doppler mode.

DETAILED DESCRIPTION:
Nipple Sparing Mastectomy (NSM) has been increasingly utilized over the last ten years for risk-reducing surgery and surgical treatment for breast cancer. The oncologic safety has been well established in multiple studies in appropriately selected individuals. Additionally, rates of wound complications and risk factors for wound problems are well documented. The intercostal perforating vessels (IPV) have been demonstrated to provide a significant proportion of the blood supply to the nipple-areolar complex1-3. Thus, preservation of these vessels is essential to reducing ischemic necrosis of the nipple-areolar complex. We propose that localization of these vessels utilizing intra-operative ultrasound (US) will reduce ischemic necrosis complications of NSM.

Objectives

* Demonstrate that US is an effective means of localizing the IPV intraoperatively.
* Evaluate the frequency of IPV preservation with the use of US.
* Measure rate and severity of ischemic necrosis when US is utilized to preserve IPV.
* Compare observed rate with historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years of age or older
* Planned nipple sparing mastectomy

Exclusion Criteria:

* Contraindication to nipple sparing mastectomy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female subjects scheduled for nipple sparing mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Localization of the intercostal perforating vessels utilizing intra-operative ultrasound (US) will reduce ischemic necrosis complications of nipple sparing mastectomy. | At the time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Maganini, MD, Principal Investigator — Amita Health
Locations (1):
- AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Palmer JH, Taylor GI. The vascular territories of the anterior chest wall. Br J Plast Surg. 1986 Jul;39(3):287-99. doi: 10.1016/0007-1226(86)90037-8. PMID 3730674
- [Background] Lemaine V, Hoskin TL, Farley DR, Grant CS, Boughey JC, Torstenson TA, Jacobson SR, Jakub JW, Degnim AC. Introducing the SKIN score: a validated scoring system to assess severity of mastectomy skin flap necrosis. Ann Surg Oncol. 2015 Sep;22(9):2925-32. doi: 10.1245/s10434-015-4409-3. Epub 2015 Jan 30. PMID 25634782